CLINICAL TRIAL: NCT02728622
Title: A Randomized Study of Chemotherapy Versus Hormonal Treatment in Patients With Ovarian Cancer Resistant or Refractory to Platinum and Taxane
Brief Title: Chemotherapy vs Hormonal Treatment in Platinum-resistant Ovarian Cancer Resistant or Refractory to Platinum and Taxane
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSGO-OC-0101
Record Dates: First submitted 2016-03-19; First posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Cancer of the Fallopian Tube
Keywords: ovarian cancer; platinum-resistant; endocrine treatment; chemotherapy; tamoxifen
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Tamoxifen; Drug Therapy; Paclitaxel; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tamoxifen (Experimental): Tamoxifen 40 mg is given orally once daily until progression
  Interventions: Drug: Tamoxifen
- Chemotherapy (Active Comparator): Paclitaxel 80 mg/m2 is given as an 1 hour infusion every 7 days or Caelyx 40 mg/m2 is given iv, first dose over 2 hours, later doses are infused over 1 hour, administered every 4 weeks or up to a maximum dose of 550 mg/m2. Until progression
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Tamoxifen — endocrine treatment
  Arms: Tamoxifen
Drug: Chemotherapy — Paclitaxel or pegylated liposomal doxorubicin
  Other Names: paclitaxel; pegylated liposomal doxorubicin
  Arms: Chemotherapy

SUMMARY:
A randomized study of chemotherapy versus hormonal treatment in patients with ovarian cancer resistant or refractory to platinum and taxane.

DETAILED DESCRIPTION:
Patients with platinum-resistant invasive epithelial ovarian, fallopian tube or peritoneal cancer will be randomized 1:2 to either hormonal treatment with Tamoxifen 40 mg daily or chemotherapy of investigator's choice (weekly paclitaxel given as an 1 hour infusion of paclitaxel 80 mg/m2 or pegylated liposomal doxorubicin 40 mg/m2 given every 4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients with invasive epithelial ovarian, fallopian tube or peritoneal cancer, being resistant to treatment with platinum and a taxane, either given in combination or sequentially.
* Patients with clinical progression during or within 6 months after end of treatment for primary disease or relapse.
* Patients with stable disease after 6 courses of chemotherapy for primary disease or relapse if further treatment is indicated.
* Patients with doubling of s-CA 125 to at least 70 IU/Ml within 3 months after end of treatment for primary disease or relapse.
* Age must be at least 18 years.
* Performance status must be 0-2 (WHO/ECOG, appendix 1).
* Informed consent given according to ICH/EU GCP guidelines and local or national laws

Exclusion Criteria:

* Patients with symptomatic brain metastasis
* Bilirubin greater than 2 x UNL (upper normal limits), white blood cell count below 3.0 x 109/L, neutrophil count below 1.5 x 109/L, platelets count below 100 x 109/L.
* Active infection or other serious underlying medical condition which might prevent the patient from receiving treatment or to be followed.
* Pregnant, lactating, or child bearing potential patients without adequate contraception
* Previous treatment with Tamoxifen.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2002-03; Primary Completion 2008-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Quality-adjusted survival | through completion of study, on average 1 year

SECONDARY OUTCOMES:
progression-free survival | through completion of study, on average 3 months
  time to progressive disease or death
overall survival | through completion of study, on average 1 year
  time to death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar B Kristensen, Prof, Study Chair — The Norwegian Radium Hospital, Oslo University Hospital

IPD SHARING:
Plan to Share IPD: No